CLINICAL TRIAL: NCT06111430
Title: The Ambidirectional Cohort Study of Neurovascular Complications After Radiation Therapy in Head and Neck Cancer Patients
Brief Title: Long-term Neurovascular Complications After Radiation Therapy in Head and Neck Cancer
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202200464B0
Record Dates: First submitted 2023-10-17; First posted 2023-11-01 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-04

CONDITIONS: Radiation Treatment; Neurovascular Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Head and neck cancer is a group of cancers develop from the soft tissues, salivary gland, mucosa of the upper respiratory or digestive system covering the oral and nasal cavity. Radiotherapy is usually the standard treatment of Head and neck cancers. In the present study, investigators aim to study the prevalence of cervical-cranial vascular complications during the early stages in these Head and neck cancer patients receiving Radiotherapy. Investigators will also compare the results between Nasopharyngeal cancer and other Head and neck cancerpatients receiving Radiotherapy.

ELIGIBILITY:
Population: Prospective cohort

Inclusion Criteria:

1. Age ≥20 years.
2. Head and neck cancer patient .
3. Had ever received radiation therapy (RT) ≦ 72 months before inclusion in the registry.
4. Had ≥ 1 brain images and cervical-cranial vascular studies between the end of RT and d date of enrolment.

Exclusion Criteria:

1. Age <20 years.
2. Patients not willing to sign the informed consent.

Population: Retrospective validation cohort

Inclusion Criteria:

1. Age ≥20 years.
2. Head and neck cancer patient.
3. Had ever received radiation therapy (RT) > 120 months before the adoption date of IRB at the participant site.
4. Had ≥ 2 brain images and cervical-cranial vascular studies between the end of RT and 6~10 years after RT, one within 5 years after RT, the other after 5 years after RT.

Exclusion Criteria:

1.Age <20 years.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise Head and neck cancer patients recruited in the prospective and retrospective cohorts. The Head and neck cancer patients in this study indicates those coded with ICD 10 (C00-13, C30-32). The coordinating center (Linkou medical center) will establish periodic communications through email and newsletters with participating sites (Keelung branch, Chia-yi branch, and etc.) to ensure data completeness and reduce the odds of loss-to follow-up of patients. We will aim to minimize data queries as much as possible, by prioritizing the completeness of the most relevant data for evaluating the main registry outcomes. We plan to follow up the patients until after 120 months after radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Significant CAS at internal carotid artery or common carotid artery | 1 year
  We define significant CAS as (a) >50% stenosis on the B-mode with peak systolic velocities ≥120 cm/s based on the hemodynamic criteria at any internal carotid artery or common carotid artery in the CDU study according to the standard ultrasound criteria35; or (b) > 50% diameter stenosis on the follow up CT or MR images.
Cerebral infarctions (CI) | 1 year
  The CI is defined whenever there were symptomatic IS occurrence of presence of asymptomatic IS on the reviewed brain MRIs.
Significant extracranial vertebral artery stenosis (VAS) | 1 year
  > 50% diameter stenosis on the follow up CT or MR images.
Significant intracranial artery stenosis | 1 year
  Presence of > 50% stenosis at intracranial ICA/VA, basilar artery, middle cerebral artery, anterior cerebral artery, or anterior cerebral artery.
Presence of carotid blow-out syndrome | 1 year
  Carotid blow out syndrome was categorized as type 1 (threaten type), type 2 (impending blowouts), and type 3 (acute CBS hemorrhage).
Presence of TLN | 1 year
  We will identify white matter lesions, contrast-enhanced lesions, Cysts, and local mass effect. The white matter lesions in the temporal lobe will be divided into three groups: mild (small focal areas), moderate (larger confluent areas) and severe (large confluent areas extending outside the radiation field with or without local mass effect). The cysts will be evaluated for size and number. The local mass effect will be classified as mild (affecting only the temporal lobe sulci), moderate (affecting the sulci and ventricles) and severe (affecting the midline of the brain).
Presence of hypothyroidism | 1 year
  Clinical hypothyroidism was diagnosed when a patient had free T4 ≤ 0.80 ng/dL with elevated TSH (>5.0 mU/L).
Tumor recurrence | 1 year
  Relapse
Mortality | 1 year
  Death

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Jiang JL, Chang JT, Huang BS, Chang TY, Sung PS, Wei YC, Lin CY, Yeh CH, Fan KH, Liu CH. Post-irradiation vertebral and carotid stenosis heightens stroke risk in head and neck cancer. BMC Cancer. 2025 Feb 11;25(1):235. doi: 10.1186/s12885-025-13647-6. PMID 39934712